CLINICAL TRIAL: NCT00849056
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Multicenter Study to Determine the Efficacy and Safety of Albiglutide When Used in Combination With Pioglitazone With or Without Metformin in Subjects With Type 2 Diabetes Mellitus
Brief Title: Safety and Efficacy of Albiglutide in Type 2 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 112755
Record Dates: First submitted 2009-02-19; First posted 2009-02-23 (Estimated); Results first posted 2014-07-01 (Estimated); Last update posted 2017-01-09 (Estimated); Status verified 2016-11

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — rGLP-1 protein

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- placebo + pioglitazone (with or without metformin) (Placebo Comparator): Placebo albiglutide weekly injection + pioglitazone (with or without metformin)
  Interventions: Drug: placebo
- albiglutide + pioglitazone (with or without metformin) (Experimental): albiglutide weekly injection + pioglitazone (with or without meformin)
  Interventions: Biological: albiglutide

INTERVENTIONS:
Biological: albiglutide — albiglutide weekly subcutaneous injection
  Arms: albiglutide + pioglitazone (with or without metformin)
Drug: placebo — placebo weekly subcutaneous injection
  Arms: placebo + pioglitazone (with or without metformin)

SUMMARY:
The purpose of this study is to determine the safety, tolerability and efficacy of albiglutide in the treatment of type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* type 2 diabetes
* BMI 20-45kg/m2

Exclusion Criteria:

* NYHA Class II to IV heart failure
* females who are pregnant, lactating, or less than 6 weeks post-partum

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 310 (Actual)
Dates: Start 2009-01; Primary Completion 2011-11 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (274):
- United States (253):
  - GSK Investigational Site, Alabaster, Alabama
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, Dothan, Alabama
  - GSK Investigational Site, Hueytown, Alabama
  - GSK Investigational Site, Mobile, Alabama
  - GSK Investigational Site, Tuscaloosa, Alabama
  - GSK Investigational Site, Chandler, Arizona
  - GSK Investigational Site, Gilbert, Arizona
  - GSK Investigational Site, Green Valley, Arizona
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, Tucson, Arizona
  - GSK Investigational Site, Bull Shoals, Arkansas
  - GSK Investigational Site, Harrisburg, Arkansas
  - GSK Investigational Site, Hot Springs, Arkansas
  - GSK Investigational Site, Jonesboro, Arkansas
  - GSK Investigational Site, Little Rock, Arkansas
  - GSK Investigational Site, Searcy, Arkansas
  - GSK Investigational Site, Buena Park, California
  - GSK Investigational Site, Carmichael, California
  - GSK Investigational Site, Chula Vista, California
  - GSK Investigational Site, Foothill Ranch, California
  - GSK Investigational Site, Fountain Valley, California
  - GSK Investigational Site, Fresno, California
  - GSK Investigational Site, Fullerton, California
  - GSK Investigational Site, Huntington Beach, California
  - GSK Investigational Site, Indio, California
  - GSK Investigational Site, Irvine, California
  - GSK Investigational Site, La Jolla, California
  - GSK Investigational Site, Lakewood, California
  - GSK Investigational Site, Long Beach, California
  - GSK Investigational Site, Los Alamitos, California
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Mission Viejo, California
  - GSK Investigational Site, Northridge, California
  - GSK Investigational Site, Palm Desert, California
  - GSK Investigational Site, Palm Springs, California
  - GSK Investigational Site, Pasadena, California
  - GSK Investigational Site, Poway, California
  - GSK Investigational Site, Riverside, California
  - GSK Investigational Site, Sacramento, California
  - GSK Investigational Site, San Diego, California
  - GSK Investigational Site, Satna Monica, California
  - GSK Investigational Site, Tarzana, California
  - GSK Investigational Site, Torrance, California
  - GSK Investigational Site, Tustin, California
  - GSK Investigational Site, Victorville, California
  - GSK Investigational Site, Walnut Creek, California
  - GSK Investigational Site, West Hills, California
  - GSK Investigational Site, Arvada, Colorado
  - GSK Investigational Site, Denver, Colorado
  - GSK Investigational Site, New Britain, Connecticut
  - GSK Investigational Site, Trumbull, Connecticut
  - GSK Investigational Site, Waterbury, Connecticut
  - GSK Investigational Site, Middletown, Delaware
  - GSK Investigational Site, Clearwater, Florida
  - GSK Investigational Site, Cocoa, Florida
  - GSK Investigational Site, Cutler Bay, Florida
  - GSK Investigational Site, Deerfield Beach, Florida
  - GSK Investigational Site, Delray Beach, Florida
  - GSK Investigational Site, Edgewater, Florida
  - GSK Investigational Site, Fort Lauderdale, Florida
  - GSK Investigational Site, Gainesville, Florida
  - GSK Investigational Site, Hallandale, Florida
  - GSK Investigational Site, Hialeah, Florida
  - GSK Investigational Site, Hollywood, Florida
  - GSK Investigational Site, Jacksonville, Florida
  - GSK Investigational Site, Lauderdale Lakes, Florida
  - GSK Investigational Site, Marianna, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, North Miami, Florida
  - GSK Investigational Site, Ocala, Florida
  - GSK Investigational Site, Orlando, Florida
  - GSK Investigational Site, Ormond Beach, Florida
  - GSK Investigational Site, Oviedo, Florida
  - GSK Investigational Site, Panama City, Florida
  - GSK Investigational Site, Pembroke Pines, Florida
  - GSK Investigational Site, Plantation, Florida
  - GSK Investigational Site, Ponte Verda, Florida
  - GSK Investigational Site, Saint Cloud, Florida
  - GSK Investigational Site, Tampa, Florida
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Blue Ridge, Georgia
  - GSK Investigational Site, Columbus, Georgia
  - GSK Investigational Site, Decatur, Georgia
  - GSK Investigational Site, Savannah, Georgia
  - GSK Investigational Site, Snellville, Georgia
  - GSK Investigational Site, Stone Mountain, Georgia
  - GSK Investigational Site, Tucker, Georgia
  - GSK Investigational Site, Honolulu, Hawaii
  - GSK Investigational Site, Boise, Idaho
  - GSK Investigational Site, Idaho Falls, Idaho
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, Evergreen Park, Illinois
  - GSK Investigational Site, La Grange, Illinois
  - GSK Investigational Site, Naperville, Illinois
  - GSK Investigational Site, Peoria, Illinois
  - GSK Investigational Site, Avon, Indiana
  - GSK Investigational Site, Evansville, Indiana
  - GSK Investigational Site, Fishers, Indiana
  - GSK Investigational Site, Indianapolis, Indiana
  - GSK Investigational Site, La Porte, Indiana
  - GSK Investigational Site, Lafayette, Indiana
  - GSK Investigational Site, South Bend, Indiana
  - GSK Investigational Site, Council Bluffs, Iowa
  - GSK Investigational Site, Des Moines, Iowa
  - GSK Investigational Site, Dubuque, Iowa
  - GSK Investigational Site, Iowa City, Iowa
  - GSK Investigational Site, Waterloo, Iowa
  - GSK Investigational Site, Arkansas City, Kansas
  - GSK Investigational Site, Mission, Kansas
  - GSK Investigational Site, Newton, Kansas
  - GSK Investigational Site, Overland Park, Kansas
  - GSK Investigational Site, Topeka, Kansas
  - GSK Investigational Site, Crescent Springs, Kentucky
  - GSK Investigational Site, Lexington, Kentucky
  - GSK Investigational Site, Louisville, Kentucky
  - GSK Investigational Site, Paducah, Kentucky
  - GSK Investigational Site, Covington, Louisiana
  - GSK Investigational Site, Lake Charles, Louisiana
  - GSK Investigational Site, Shreveport, Louisiana
  - GSK Investigational Site, Baltimore, Maryland
  - GSK Investigational Site, Hyattsville, Maryland
  - GSK Investigational Site, Oxon Hill, Maryland
  - GSK Investigational Site, Haverhill, Massachusetts
  - GSK Investigational Site, Bay City, Michigan
  - GSK Investigational Site, Benzonia, Michigan
  - GSK Investigational Site, Bloomfield Hills, Michigan
  - GSK Investigational Site, Dearborn, Michigan
  - GSK Investigational Site, Interlochen, Michigan
  - GSK Investigational Site, Kalamazoo, Michigan
  - GSK Investigational Site, Saint Clair Shores, Michigan
  - GSK Investigational Site, Minneapolis, Minnesota
  - GSK Investigational Site, Gulfport, Mississippi
  - GSK Investigational Site, Picayune, Mississippi
  - GSK Investigational Site, Rolling Fork, Mississippi
  - GSK Investigational Site, Chesterfield, Missouri
  - GSK Investigational Site, Jefferson City, Missouri
  - GSK Investigational Site, Kansas City, Missouri
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, West Plains, Missouri
  - GSK Investigational Site, Billings, Montana
  - GSK Investigational Site, Butte, Montana
  - GSK Investigational Site, Great Falls, Montana
  - GSK Investigational Site, Broken Bow, Nebraska
  - GSK Investigational Site, Lincoln, Nebraska
  - GSK Investigational Site, Omaha, Nebraska
  - GSK Investigational Site, Las Vegas, Nevada
  - GSK Investigational Site, Berlin, New Jersey
  - GSK Investigational Site, Elizabeth, New Jersey
  - GSK Investigational Site, Haddon Heights, New Jersey
  - GSK Investigational Site, Hainesport, New Jersey
  - GSK Investigational Site, Stratford, New Jersey
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, North Massapequa, New York
  - GSK Investigational Site, Asheboro, North Carolina
  - GSK Investigational Site, Asheville, North Carolina
  - GSK Investigational Site, Burlington, North Carolina
  - GSK Investigational Site, Calabash, North Carolina
  - GSK Investigational Site, Chadbourn, North Carolina
  - GSK Investigational Site, Durham, North Carolina
  - GSK Investigational Site, Fayetteville, North Carolina
  - GSK Investigational Site, Greensboro, North Carolina
  - GSK Investigational Site, Hickory, North Carolina
  - GSK Investigational Site, Lenoir, North Carolina
  - GSK Investigational Site, Mint Hill, North Carolina
  - GSK Investigational Site, Morehead City, North Carolina
  - GSK Investigational Site, Shelby, North Carolina
  - GSK Investigational Site, Tabor City, North Carolina
  - GSK Investigational Site, Akron, Ohio
  - GSK Investigational Site, Canal Fulton, Ohio
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Cleveland, Ohio
  - GSK Investigational Site, Columbus, Ohio
  - GSK Investigational Site, Dayton, Ohio
  - GSK Investigational Site, Kettering, Ohio
  - GSK Investigational Site, Mason, Ohio
  - GSK Investigational Site, Maumee, Ohio
  - GSK Investigational Site, Thornville, Ohio
  - GSK Investigational Site, Zanesville, Ohio
  - GSK Investigational Site, Oklahoma City, Oklahoma
  - GSK Investigational Site, Tulsa, Oklahoma
  - GSK Investigational Site, Ashland, Oregon
  - GSK Investigational Site, Bensalem, Pennsylvania
  - GSK Investigational Site, Carlisle, Pennsylvania
  - GSK Investigational Site, Downington, Pennsylvania
  - GSK Investigational Site, Feasterville, Pennsylvania
  - GSK Investigational Site, Harrisburg, Pennsylvania
  - GSK Investigational Site, Landsdale, Pennsylvania
  - GSK Investigational Site, Melrose Park, Pennsylvania
  - GSK Investigational Site, Tipton, Pennsylvania
  - GSK Investigational Site, Uniontown, Pennsylvania
  - GSK Investigational Site, Cumberland, Rhode Island
  - GSK Investigational Site, East Providence, Rhode Island
  - GSK Investigational Site, Columbia, South Carolina
  - GSK Investigational Site, Greenville, South Carolina
  - GSK Investigational Site, Greer, South Carolina
  - GSK Investigational Site, Murrells Inlet, South Carolina
  - GSK Investigational Site, North Myrtle Beach, South Carolina
  - GSK Investigational Site, Orangeburg, South Carolina
  - GSK Investigational Site, Simpsonville, South Carolina
  - GSK Investigational Site, Bristol, Tennessee
  - GSK Investigational Site, Chattanooga, Tennessee
  - GSK Investigational Site, Clarksville, Tennessee
  - GSK Investigational Site, Columbia, Tennessee
  - GSK Investigational Site, Crossville, Tennessee
  - GSK Investigational Site, Fayetteville, Tennessee
  - GSK Investigational Site, Germantown, Tennessee
  - GSK Investigational Site, Johnson City, Tennessee
  - GSK Investigational Site, McKenzie, Tennessee
  - GSK Investigational Site, Memphis, Tennessee
  - GSK Investigational Site, Nashville, Tennessee
  - GSK Investigational Site, Tullahoma, Tennessee
  - GSK Investigational Site, Arlington, Texas
  - GSK Investigational Site, Bedford, Texas
  - GSK Investigational Site, Cleburne, Texas
  - GSK Investigational Site, Corpus Christi, Texas
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Deer Park, Texas
  - GSK Investigational Site, El Paso, Texas
  - GSK Investigational Site, Fort Worth, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Hurst, Texas
  - GSK Investigational Site, Katy, Texas
  - GSK Investigational Site, Lake Jackson, Texas
  - GSK Investigational Site, Lewisville, Texas
  - GSK Investigational Site, Midland, Texas
  - GSK Investigational Site, North Richland Hills, Texas
  - GSK Investigational Site, Odessa, Texas
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Schertz, Texas
  - GSK Investigational Site, Sugar Land, Texas
  - GSK Investigational Site, Sugarland, Texas
  - GSK Investigational Site, Bountiful, Utah
  - GSK Investigational Site, Orem, Utah
  - GSK Investigational Site, Salt Lake City, Utah
  - GSK Investigational Site, West Jordan, Utah
  - GSK Investigational Site, West Valley City, Utah
  - GSK Investigational Site, South Burlington, Vermont
  - GSK Investigational Site, Burke, Virginia
  - GSK Investigational Site, Hampton, Virginia
  - GSK Investigational Site, Manassas, Virginia
  - GSK Investigational Site, Norfolk, Virginia
  - GSK Investigational Site, Richmond, Virginia
  - GSK Investigational Site, Suffolk, Virginia
  - GSK Investigational Site, Weber City, Virginia
  - GSK Investigational Site, Federal Way, Washington
  - GSK Investigational Site, Renton, Washington
  - GSK Investigational Site, Richland, Washington
  - GSK Investigational Site, Selah, Washington
  - GSK Investigational Site, Spokane, Washington
  - GSK Investigational Site, Tacoma, Washington
  - GSK Investigational Site, Lewisburg, West Virginia
  - GSK Investigational Site, Milwaukee, Wisconsin
- India (2):
  - GSK Investigational Site, Aurangabad
  - GSK Investigational Site, Pune
- Peru (5):
  - GSK Investigational Site, Arequipa, Arequipa
  - GSK Investigational Site, Lima, Lima Province
  - GSK Investigational Site, El Agustino, Lima region
  - GSK Investigational Site, Huacho, Lima region
  - GSK Investigational Site, Trujillo
- South Africa (4):
  - GSK Investigational Site, Port Elizabeth, Eastern Cape
  - GSK Investigational Site, Phoenix, KwaZulu-Natal
  - GSK Investigational Site, Kempton Park
  - GSK Investigational Site, Somerset West
- South Korea (2):
  - GSK Investigational Site, Seongnam-si
  - GSK Investigational Site, Suwon, Kyonggi-do
- United Kingdom (8):
  - GSK Investigational Site, Canterbury, Kent
  - GSK Investigational Site, Blackpool, Lancashire
  - GSK Investigational Site, Sunbury-on-Thames, Middlesex
  - GSK Investigational Site, Port Glasgow, Renfrewshire
  - GSK Investigational Site, Coventry, West Midlands
  - GSK Investigational Site, Glasgow
  - GSK Investigational Site, Liverpool
  - GSK Investigational Site, London

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Home PD, Ahren B, Reusch JEB, Rendell M, Weissman PN, Cirkel DT, Miller D, Ambery P, Carr MC, Nauck MA. Three-year data from 5 HARMONY phase 3 clinical trials of albiglutide in type 2 diabetes mellitus: Long-term efficacy with or without rescue therapy. Diabetes Res Clin Pract. 2017 Sep;131:49-60. doi: 10.1016/j.diabres.2017.06.013. Epub 2017 Jun 15. PMID 28683300
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Individual Participant Data Set: 112755 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 112755 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 112755 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 112755 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 112755 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 112755 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 112755 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants (par.) who met eligibility criteria and completed a 4-week Run-in/Stabilization Period were then randomized to a 156-week Treatment Period, followed by 8 weeks of post-treatment follow-up. A total of 450 par. were screened; 310 par. were randomized, and 301 par. received >=1 treatment dose.
Groups:
- Placebo + Pioglitazone With or Without Metformin: Participants received matching placebo as a subcutaneous injection weekly via a fully disposable pen injector system and pioglitazone (>=30 milligrams [mg]/day, unless there was documented evidence that the participant could not tolerate that dose, in which case they were allowed 15 mg/day) with or without metformin as appropriate. Participants did not receive investigational product during the Follow-up Period.
- Albiglutide 30 mg + Pioglitazone With or Without Metformin: Participants received albiglutide 30 milligrams (mg) as a subcutaneous injection weekly via a fully disposable pen injector system and pioglitazone (>=30 mg/day, unless there was documented evidence that the participant could not tolerate that dose, in which case they were allowed 15 mg/day) with or without metformin as appropriate. Participants did not receive investigational product during the Follow-up Period.
Period: Treatment Period (TP) (156 Weeks)
Arm/Group | Placebo + Pioglitazone With or Without Metformin | Albiglutide 30 mg + Pioglitazone With or Without Metformin
Started | 151 | 150
Completed | 88 | 100
Not Completed | 63 | 50
Not completed — Adverse Event | 13 | 11
Not completed — Protocol Violation | 3 | 6
Not completed — Noncompliance | 3 | 3
Not completed — Lost to Follow-up | 7 | 5
Not completed — Withdrawal by Subject | 31 | 18
Not completed — Physician Decision | 3 | 3
Not completed — Termination of Study/Site by GSK | 1 | 4
Not completed — Calcitonin Out of Range | 1 | 0
Not completed — Pregnancy | 1 | 0
Period: Follow-up Period (FUP) (8 Weeks)
Arm/Group | Placebo + Pioglitazone With or Without Metformin | Albiglutide 30 mg + Pioglitazone With or Without Metformin
Started | 149 (Par. withdrawing from the TP could enter the FUP. Two par. did not participate in the FUP.) | 149 (Par. withdrawing from the TP could enter the FUP. One par. did not participate in the FUP.)
Completed | 122 | 124
Not Completed | 27 | 25
Not completed — Adverse Event | 1 | 3
Not completed — Noncompliance | 0 | 1
Not completed — Lost to Follow-up | 14 | 9
Not completed — Withdrawal by Subject | 9 | 7
Not completed — Physician Decision | 1 | 1
Not completed — Termination of Study/Site by GSK | 1 | 4
Not completed — Early Termination | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo + Pioglitazone With or Without Metformin | Albiglutide 30 mg + Pioglitazone With or Without Metformin | Total
Number analyzed (Participants) | 151 | 150 | 301
Age, Continuous [Mean (Standard Deviation); unit: Years] | 54.9 (9.40) | 55.2 (9.98) | 55.0 (9.67)
Gender [Count of Participants; unit: Participants]
  Female | 63 | 58 | 121
  Male | 88 | 92 | 180
Race/Ethnicity, Customized [Number; unit: Participants]
  African American/African Heritage | 20 | 19 | 39
  American Indian or Alaskan Native | 15 | 18 | 33
  Asian - Central/South Asian Heritage | 1 | 2 | 3
  Asian - East Asian Heritage | 2 | 3 | 5
  Asian - Japanese Heritage | 1 | 1 | 2
  Asian - South East Asian Heritage | 2 | 0 | 2
  Native Hawaiian or other Pacific Islander | 2 | 1 | 3
  White - Arabic/North African Heritage | 2 | 2 | 4
  White - White/Caucasian/European Heritage | 106 | 104 | 210

OUTCOME MEASURES:

1. Secondary Outcome: Change From Baseline in HbA1c at Weeks 104 and 156
Description: HbA1c is a form of hemoglobin that is measured primarily to identify the average plasma glucose concentration over a 2- to 3-month period. Baseline HbA1c value is defined as the last non-missing value before the start of treatment. Change from Baseline was calculated as the post-Baseline value minus the Baseline value. This analysis used observed HbA1c values, excluding those obtained after hyperglycemia rescue; no missing data imputation was performed.
Time Frame: Baseline and Weeks 104 and 156
Population: ITT Population with observed values. Only those participants with a value at Baseline and at the specified visit were analyzed (represented by n=X, X in the category titles).
Measure: Mean (Standard Deviation); unit: Percentage of HbA1c in the blood
Arm/Group | Placebo + Pioglitazone With or Without Metformin | Albiglutide 30 mg + Pioglitazone With or Without Metformin
Number analyzed (Participants) | 29 | 72
Percentage of HbA1c in the blood
  Week 104, n= 29, 72 | -0.72 (0.845) | -0.92 (1.038)
  Week 156, n=26, 54 | -0.50 (0.805) | -0.87 (0.926)

2. Primary Outcome: Change From Baseline (BL) in Glycosylated Hemoglobin (HbA1c) at Week 52
Description: HbA1c is a form of hemoglobin that is measured primarily to identify the average plasma glucose concentration over a 2- to 3-month period. The BL HbA1c value is defined as the last non-missing value before the start of treatment. Change from BL was calculated as the value at Week 52 minus the value at BL. Based on analysis of covariance (ANCOVA): change = treatment + BL HbA1c + prior myocardial infarction history + age category + region + current antidiabetic therapy. The last observation carried forward (LOCF) method was used to impute missing post-BL HbA1c values; the last non-missing post-BL on-treatment measurement was used to impute the missing measurement. HbA1c values obtained after hyperglycemic rescue were treated as missing and were replaced with pre-rescue values. One Intent-to-Treat (ITT) participant (par.) had all post-BL HbA1c measurements occur after hyperglycemic rescue. This par. is included in the ITT Population counts but did not contribute to this analysis.
Time Frame: Baseline and Week 52
Population: Intent-to-Treat (ITT) Population with LOCF: all randomized par. who received >=1 dose of study medication and who had a BL assessment and >=1 post-BL assessment of HbA1c. Only par. with a value at BL and at the specified visit were analyzed. Values were carried forward for par. who were rescued or discontinued from active treatment before Week 52.
Measure: Least Squares Mean (Standard Error); unit: Percentage of HbA1c in the blood
Arm/Group | Placebo + Pioglitazone With or Without Metformin | Albiglutide 30 mg + Pioglitazone With or Without Metformin
Number analyzed (Participants) | 149 | 149
Percentage of HbA1c in the blood | -0.05 (0.071) | -0.81 (0.071)
Statistical Analysis 1: Comparison: Placebo + Pioglitazone With or Without Metformin vs Albiglutide 30 mg + Pioglitazone With or Without Metformin; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Net) = -0.75, 95% CI 2-sided [-0.95 to -0.56]

3. Secondary Outcome: Time to Hyperglycemia Rescue
Description: Participants who experienced persistent hyperglycemia (high blood glucose) could have qualified for hyperglycemia rescue. The conditions for hyperglycemia rescue were as follows: FPG >=280 milligrams/deciliter (mg/dL) between >=Week 2 and <Week 4; FPG >=250 mg/dL between >=Week 4 and <Week 12; HbA1c >=8.5% and a <=0.5% reduction from Baseline between >=Week 12 and <Week 24; HbA1c >=8.5% between >=Week 24 and <Week 48; HbA1c >=8.0% between >= Week 48 and <Week 156. Participants could have been rescued at any time on or after Week 2. Time to hyperglycemia rescue is defined as the time between the date of the first dose of study medication and the date of hyperglycemia rescue plus 1 day, or the time between the date of the first dose of study medication and the date of the last visit during the active treatment period plus 1 day for participants not requiring rescue. This time was divided by 7 to express the result in weeks.
Time Frame: From the start of study medication until the end of the treatment (up to Week 156)
Population: ITT Population. Only those participants with a value at Baseline and at the specified visit were analyzed.
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Placebo + Pioglitazone With or Without Metformin | Albiglutide 30 mg + Pioglitazone With or Without Metformin
Number analyzed (Participants) | 149 | 150
Weeks | 52.86 (0.674) [48.86 to 79.43] | NA (0.812) [NA to NA] — There were too few events of hyperglycemia rescue (<50% of participants with events) to calculate the median and confidence interval.

4. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG) at Week 52
Description: The FPG test measures blood sugar levels after the participant has not eaten (fasted) for 12 to 14 hours. The Baseline FPG value is the last non-missing value before the start of treatment. The LOCF method was used to impute missing post-Baseline FPG values. FPG values obtained after hyperglycemia rescue were treated as missing and replaced with pre-rescue values. Change from Baseline was calculated as the post-Baseline value minus the Baseline value. Based on ANCOVA: change = treatment + Baseline weight + prior myocardial infarction history + age category + region + current antidiabetic therapy.
Time Frame: Baseline and Week 52
Population: Intent-to-Treat (ITT) Population with LOCF. Only those participants with a value at Baseline and at the specified visit were analyzed. Values were carried forward for participants who were rescued or discontinued from active treatment before Week 52.
Measure: Least Squares Mean (Standard Error); unit: Millimoles per liter (mmol/L)
Arm/Group | Placebo + Pioglitazone With or Without Metformin | Albiglutide 30 mg + Pioglitazone With or Without Metformin
Number analyzed (Participants) | 149 | 149
Millimoles per liter (mmol/L) | 0.35 (0.197) | -1.28 (0.197)

5. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG) at Week 156
Description: The Baseline FPG value is the last non-missing value before the start of treatment. Change from Baseline was calculated as the post-Baseline FPG minus the Baseline FPG.
Time Frame: Baseline and Week 156
Population: ITT Population with observed values. Only those participants with a value at Baseline and at the specified visit were analyzed. This analysis used observed FPG values excluding those obtained after hyperglycemia rescue; no missing data imputation was performed.
Measure: Mean (Standard Deviation); unit: Millimoles per liter (mmol/L)
Arm/Group | Placebo + Pioglitazone With or Without Metformin | Albiglutide 30 mg + Pioglitazone With or Without Metformin
Number analyzed (Participants) | 25 | 54
Millimoles per liter (mmol/L) | 0.03 (1.950) | -1.26 (1.476)

6. Secondary Outcome: Number of Participants Who Achieved Clinically Meaningful HbA1c Response Levels of <6.5%, <7%, and <7.5% at Week 52
Description: The number of participants who achieved the HbA1c treatment goal (i.e., HbA1c response levels of <6.5%, <6.5%, and <7.0% at Week 52) were assessed.
Time Frame: Week 52
Population: ITT Population with LOCF. Only those participants with a value at Baseline and at the specified visit were analyzed. Values were carried forward for participants who were rescued or discontinued from active treatment before Week 52.
Measure: Number; unit: Participants
Arm/Group | Placebo + Pioglitazone With or Without Metformin | Albiglutide 30 mg + Pioglitazone With or Without Metformin
Number analyzed (Participants) | 149 | 149
Participants
  HbA1c <6.5% | 8 | 37
  HbA1c <7% | 22 | 66
  HbA1c <7.5% | 44 | 96

7. Secondary Outcome: Number of Participants Who Achieved Clinically Meaningful HbA1c Response Levels of <6.5%, <7%, and <7.5% at Week 156
Description: The number of participants who achieved the HbA1c treatment goal (i.e., HbA1c response levels of <6.5%, <6.5%, and <7.0% at Week 156) were assessed.
Time Frame: Week 156
Population: ITT Population with observed values. Only those participants with a value at Baseline and at the specified visit were analyzed. This analysis used observed HbA1c values excluding those obtained after hyperglycemia rescue; no missing data imputation was performed.
Measure: Number; unit: Participants
Arm/Group | Placebo + Pioglitazone With or Without Metformin | Albiglutide 30 mg + Pioglitazone With or Without Metformin
Number analyzed (Participants) | 26 | 54
Participants
  HbA1c <6.5% | 7 | 20
  HbA1c <7% | 12 | 32
  HbA1c <7.5% | 17 | 44

8. Secondary Outcome: Change From Baseline in Body Weight at Week 52
Description: The Baseline value is the last non-missing value before the start of treatment. Change from Baseline was calculated as the post-Baseline weight minus the Baseline weight. The LOCF method was used to impute missing post-Baseline weight values. Weight values obtained after hyperglycemia rescue were treated as missing and replaced with prerescue values. Based on ANCOVA: change = treatment + Baseline weight + prior myocardial infarction history + age category + region + current antidiabetic therapy.
Time Frame: Baseline and Week 52
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: Kilograms
Arm/Group | Placebo + Pioglitazone With or Without Metformin | Albiglutide 30 mg + Pioglitazone With or Without Metformin
Number analyzed (Participants) | 149 | 149
Kilograms | 0.45 (0.348) | 0.28 (0.348)

9. Secondary Outcome: Change From Baseline in Body Weight at Week 156
Description: The Baseline value is the last non-missing value before the start of treatment. Change from Baseline was calculated as the post-Baseline weight minus the Baseline weight.
Time Frame: Baseline and Week 156
Population: ITT Population with observed values. Only those participants who were available at the indicated time points were analyzed. This analysis used observed body weight values excluding those obtained after hyperglycemia rescue; no missing data imputation was performed.
Measure: Mean (Standard Deviation); unit: Kilograms
Arm/Group | Placebo + Pioglitazone With or Without Metformin | Albiglutide 30 mg + Pioglitazone With or Without Metformin
Number analyzed (Participants) | 26 | 55
Kilograms | 1.50 (6.939) | -0.16 (6.284)

ADVERSE EVENTS:
Time Frame: On-treatment serious adverse events (SAEs) and non-serious AEs, defined as those events that had a start date on or after the first day of study medication and within 56 days after the end of study medication (up to Week 156), are reported.
Description: SAEs and non-serious AEs are reported for members of the Safety Population, comprised of all participants who received at least one dose of study treatment.
Arm/Group | Placebo + Pioglitazone With or Without Metformin | Albiglutide 30 mg + Pioglitazone With or Without Metformin
Serious Adverse Events (participants affected / at risk) | 28/151 | 15/150
Other Adverse Events (participants affected / at risk) | 117/151 | 126/150
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo + Pioglitazone With or Without Metformin (N=151) | Albiglutide 30 mg + Pioglitazone With or Without Metformin (N=150)
Coronary artery disease (Cardiac disorders) | 2 | 2
Acute myocardial infarction (Cardiac disorders) | 0 | 2
Angina unstable (Cardiac disorders) | 0 | 1
Aortic valve incompetence (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 1 | 0
Cardiomyopathy (Cardiac disorders) | 1 | 0
Coronary artery stenosis (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0
Sick sinus syndrome (Cardiac disorders) | 1 | 0
Cellulitis (Infections and infestations) | 2 | 1
Abscess limb (Infections and infestations) | 1 | 1
Pneumonia (Infections and infestations) | 0 | 2
Appendicitis perforated (Infections and infestations) | 0 | 1
Diverticulitis (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 1 | 0
Viral infection (Infections and infestations) | 0 | 1
Vulval abscess (Infections and infestations) | 1 | 0
Colonic fistula (Gastrointestinal disorders) | 0 | 1
Diabetic gastroparesis (Gastrointestinal disorders) | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Breast cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Chest pain (General disorders) | 3 | 0
Cholecystitis acute (Hepatobiliary disorders) | 2 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 1
Renal colic (Renal and urinary disorders) | 0 | 1
Renal impairment (Renal and urinary disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 2 | 0
Face injury (Injury, poisoning and procedural complications) | 1 | 0
Obesity (Metabolism and nutrition disorders) | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Major depression (Psychiatric disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo + Pioglitazone With or Without Metformin (N=151) | Albiglutide 30 mg + Pioglitazone With or Without Metformin (N=150)
Upper respiratory tract infection (Infections and infestations) | 24 | 24
Urinary tract infection (Infections and infestations) | 9 | 17
Sinusitis (Infections and infestations) | 9 | 15
Nasopharyngitis (Infections and infestations) | 22 | 12
Bronchitis (Infections and infestations) | 15 | 10
Gastroenteritis (Infections and infestations) | 2 | 7
Pharyngitis (Infections and infestations) | 7 | 6
Influenza (Infections and infestations) | 2 | 6
Cellulitis (Infections and infestations) | 4 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 13 | 15
Back pain (Musculoskeletal and connective tissue disorders) | 10 | 13
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 10 | 13
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 6 | 11
Pain in extremity (Musculoskeletal and connective tissue disorders) | 11 | 7
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 6
Neck pain (Musculoskeletal and connective tissue disorders) | 3 | 5
Muscle spasms (Musculoskeletal and connective tissue disorders) | 7 | 4
Bursitis (Musculoskeletal and connective tissue disorders) | 4 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 4 | 0
Diarrhoea (Gastrointestinal disorders) | 16 | 22
Nausea (Gastrointestinal disorders) | 18 | 18
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 9
Vomiting (Gastrointestinal disorders) | 6 | 8
Toothache (Gastrointestinal disorders) | 4 | 8
Abdominal pain upper (Gastrointestinal disorders) | 6 | 6
Constipation (Gastrointestinal disorders) | 2 | 5
Dyspepsia (Gastrointestinal disorders) | 5 | 4
Gastritis (Gastrointestinal disorders) | 3 | 4
Abdominal pain (Gastrointestinal disorders) | 8 | 2
Oedema peripheral (General disorders) | 16 | 15
Fatigue (General disorders) | 7 | 10
Injection site reaction (General disorders) | 5 | 8
Injection site haemorrhage (General disorders) | 1 | 7
Injection site haematoma (General disorders) | 4 | 6
Pyrexia (General disorders) | 4 | 3
Injection stie pruritis (General disorders) | 5 | 0
Headache (Nervous system disorders) | 18 | 13
Dizziness (Nervous system disorders) | 5 | 10
Hypoaesthesia (Nervous system disorders) | 2 | 4
Neuropathy peripheral (Nervous system disorders) | 6 | 2
Carpal tunnel syndrome (Nervous system disorders) | 6 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 13 | 25
Decreased appetite (Metabolism and nutrition disorders) | 4 | 3
Dyslipidaemia (Metabolism and nutrition disorders) | 8 | 2
Contusion (Injury, poisoning and procedural complications) | 9 | 12
Laceration (Injury, poisoning and procedural complications) | 2 | 7
Meniscus lesion (Injury, poisoning and procedural complications) | 2 | 4
Ligament sprain (Injury, poisoning and procedural complications) | 4 | 3
Procedural pain (Injury, poisoning and procedural complications) | 4 | 3
Muscle strain (Injury, poisoning and procedural complications) | 5 | 2
Limb injury (Injury, poisoning and procedural complications) | 4 | 2
Hypertension (Vascular disorders) | 15 | 17
Cough (Respiratory, thoracic and mediastinal disorders) | 8 | 10
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 4 | 8
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 | 4
Anxiety (Psychiatric disorders) | 6 | 7
Depression (Psychiatric disorders) | 5 | 4
Insomnia (Psychiatric disorders) | 4 | 4
Cataract (Eye disorders) | 3 | 7
Diabetic retinopathy (Eye disorders) | 2 | 7
Presbyopia (Eye disorders) | 4 | 2
Refraction disorder (Eye disorders) | 4 | 1
Pruritis (Skin and subcutaneous tissue disorders) | 1 | 5
Rash (Skin and subcutaneous tissue disorders) | 3 | 4
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 4
Anaemia (Blood and lymphatic system disorders) | 9 | 6
Vertigo (Ear and labyrinth disorders) | 2 | 5
Ear pain (Ear and labyrinth disorders) | 4 | 1
Seasonal allergy (Immune system disorders) | 5 | 5
Nephrolithiasis (Renal and urinary disorders) | 2 | 5
Renal cyst (Renal and urinary disorders) | 4 | 0
Palpitations (Cardiac disorders) | 0 | 4
Angina pectoris (Cardiac disorders) | 4 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.